CLINICAL TRIAL: NCT04318041
Title: Evaluation of the Structural Modification Effect of Diacerein (Artrodar®) in Knee Osteoarthritic Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAR-THA-19-01
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, hospital pharmacists and monitors are blind to the treatment. The analysis of the results will be performed blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diacerein (Artrodar) (Experimental)
  Interventions: Drug: Artrodar
- placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Artrodar — Diacerein (Artrodar):
  D1-D28 (1 month): Artrodar (50 mg) 1 x 1 with evening meal D29-end of study (23 months): Artrodar (50 mg) 1 x 2 with meal
  Arms: diacerein (Artrodar)
Drug: Placebos — Placebo:
  D1-D28 (1 month): Placebo 1 x 1 with evening meal D29-end of study (23 months) Placebo 1 x 2 with meal
  Arms: placebo

SUMMARY:
This study evaluates the structure-modifying effect of Diacerein (Artrodar ®) in knee osteoarthritic (OA) patients by measuring total cartilage volume from magnetic resonance imaging (MRI) of the knee. Half of participants will receive Diacerein (Artrodar ®), while the other half will receive a placebo.

DETAILED DESCRIPTION:
Diacerein (Artrodar ®) participants take 1x1 with evening meal for 1 month (D1-D28) then 1x2 with morning and evening meal for 23 months (D29-end of study). Placebo participants take 1x1 with evening meal for 1 month (D1-D28) then 1x2 with morning and evening meal for 23 months (D29-end of study).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 40 and 65 years who diagnosed with primary OA knee (medial tibiofemoral compartment) according to ACR criteria
2. Grade II-III OA severity that classified by the Kellgren-Lawrence classification
3. Varus malalignment ≤ 15°
4. Body mass index (BMI) ≤ 30 kg/m2
5. Pain on walking at 15 metres ≥ 30 mm using 100 mm visual analogue pain score (VAPS)
6. Evidence of adequate contraceptive methods in women of childbearing age

Exclusion Criteria:

1. Accompanying osteoarthritis of the hip of sufficient severity to interfere with the functional assessment of the knee
2. Intra-articular treatment with any product (corticosteroids in the last 3 months, glycosaminoglycans, hyaluronic acid in the last 6 months, etc.), joint lavage or arthroscopic procedures within 6 months before the start of the study
3. Oral corticosteroids, oral symptomatic slow acting drug for OA (SYSADOA) treatment (chondroitin sulfate, glucosamine sulfate, piascledin, diacerein) within last 3 months
4. Current treatment with anti-depressants, tranquilisers, antacids or antibiotics
5. Poor general health or other conditions which would make regular hospital attendance difficult
6. Primary inflammatory painful conditions of the knee (e.g. rheumatoid arthritis, psoriatic arthropathy, pseudo-gout)
7. Painful knee conditions other than osteoarthritis (e.g. Sudeck's atrophy, intra-articular neoplasm, villonodular synovitis)
8. Evolving arthritis requiring surgery within the coming year;
9. Persistent diarrhoea (> 3 stools /24 h) or laxative use (any laxative use is to be stopped before inclusion in the trial)
10. Severe gastrointestinal disorders, indications or history of severe gastrointestinal disorders (e.g. gastric or duodenal ulcers, ulcerative colitis, Crohn's syndrome, diverticulitis, recurrent pancreatitis)
11. Renal insufficiency (estimate glomerular filtration rate ≤ 60 ml/min/1.73 m2)
12. Hepatic disease (transaminases > 2.5 x upper limit of normal values (ULN) or total bilirubin > 2 x ULN) or history of alcoholism and liver disease
13. Severe parenchymal organ disease
14. History of heart attack or stroke, or have had serious diseases of the heart such as congestive heart failure, or taking clopidogrel.
15. Patient with diabetes mellitus (DM) who has heamoglobin A1c level > 8%
16. Patient with hypertension who has systolic blood pressure > 150 mmHg or diastolic Blood pressure > 95 mmHg
17. Pregnancy or lactation
18. Participation in a drug clinical trial within the 3 months before the start of the study;
19. Ascertained hypersensitivity to the active ingredient diacerein, to similar compounds, to the excipients or to paracetamol, naproxen, and omeprazole
20. Contraindications for magnetic resonance imaging (MRI) assessment such as heart pacemaker, aneurysm clip or claustrophobia
21. Knee size measured at lower thigh > 50 cm

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-11-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cartilage volume measured by MRI of the affected knee. | Change from Day 0 cartilage volume at Day 336, Day 672
  Cartilage volume in cc
Bone marrow lesions measured by MRI of the affected knee. | Change from Day 0 Bone marrow lesions at Day 336, Day 672
  Bone marrow lesions in mm3
Synovitis measured by MRI of the affected knee. | Change from Day 0 Synovial tissue volume at Day 336, Day 672
  Synovial tissue volume in mm3
Joint space width at narrowest point at medial compartment measured by X-ray (Full extension, weight-bearing position) | Change from Day -7 to -30 Joint space width at Day 168, Day 336, Day 504, Day 672
  Joint space width in mm

SECONDARY OUTCOMES:
Pain at rest | Day 0, Day 28, Day 84, Day 168, Day 252, Day 336, Day 420, Day 504, Day 588, Day 672
  Visual analogue scale (VAS) 0-100 mm. 0 is no pain, 100 is extreme pain.
Pain on walking at 15 meters | Day -7 to -30, Day 0, Day 28, Day 84, Day 168, Day 252, Day 336, Day 420, Day 504, Day 588, Day 672
  Visual analogue scale (VAS) 0-100 mm. 0 is no pain, 100 is extreme pain.
KOOs | Day 0, Day 28, Day 84, Day 168, Day 252, Day 336, Day 420, Day 504, Day 588, Day 672
  Knee and Osteoarthritis Outcome Score from 1-5 Likert scale score with higher scores denoting worse pain and disability.
EQ5D5L | Day 0, Day 28, Day 84, Day 168, Day 252, Day 336, Day 420, Day 504, Day 588, Day 672
  EQ5D5L is a standardized instrument for measuring generic health status
Time up-and-go test | Day 0, Day 28, Day 84, Day 168, Day 252, Day 336, Day 420, Day 504, Day 588, Day 672
Physician and Patient's global assessment | Day 168, Day 336, Day 672
  Visual analogue scale (VAS) 0-100 mm to assess efficacy and tolerability by physician and patient. 0 is not effective/ no tolerate, 100 is very effective/ very good.
Rescued medicine consumption | Day 28, Day 84, Day 168, Day 252, Day 336, Day 420, Day 504, Day 588, Day 672
Oxford Knee Questionnaire | Day 0, Day 28, Day 84, Day 168, Day 252, Day 336, Day 420, Day 504, Day 588, Day 672
  1-5 Likert scale score with higher scores denoting worse pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Nipaporn Jitsook, Study Director — TRB Chemedica
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No